CLINICAL TRIAL: NCT05002270
Title: A Phase 1/2, Multi-Center, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Evidence of Antitumor Activity of JAB-21822 Monotherapy and Combination Therapy in Adult Patients With Advanced Solid Tumors Harboring KRAS G12C Mutation
Brief Title: JAB-21822 Activity in Adult Patients With Advanced Solid Tumors Harboring KRAS G12C Mutation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jacobio Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JAB-21822-1001
Record Dates: First submitted 2021-07-26; First posted 2021-08-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor; NSCLC; CRC
Keywords: KRAS G12C Mutant Advanced Solid Tumor; NSCLC; CRC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cetuximab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A0, JAB-21822 monotherapy, Phase 1, Dose Escalation (Experimental): Dose escalation of JAB-21822 will be administered alone to determine the MTD and RP2D
  Interventions: Drug: JAB-21822 (KRAS G12C inhibitor)
- Arm A1, JAB-21822 monotherapy, Phare 2, Dose Expansion (Experimental): JAB-21822 will be administered alone at RP2D in selected cancer type patients to evaluate the preliminary antitumor activity.
  Interventions: Drug: JAB-21822 (KRAS G12C inhibitor)
- Experimental: Arm B, JAB-21822 combination with Cetuximab, Phase 2, Dose Expansion (Experimental): JAB-21822 will be administered together with Cetuximab in mCRC patients to evaluate the preliminary antitumor activity.
  Interventions: Drug: JAB-21822 (KRAS G12C inhibitor); Drug: Cetuximab (EGFR inhibitor)

INTERVENTIONS:
Drug: JAB-21822 (KRAS G12C inhibitor) — Administered orally
  Arms: Arm A0, JAB-21822 monotherapy, Phase 1, Dose Escalation
Drug: JAB-21822 (KRAS G12C inhibitor) — Administered orally
  Arms: Arm A1, JAB-21822 monotherapy, Phare 2, Dose Expansion
Drug: JAB-21822 (KRAS G12C inhibitor) — Administered orally
  Arms: Experimental: Arm B, JAB-21822 combination with Cetuximab, Phase 2, Dose Expansion
Drug: Cetuximab (EGFR inhibitor) — Administered IV
  Arms: Experimental: Arm B, JAB-21822 combination with Cetuximab, Phase 2, Dose Expansion

SUMMARY:
This study is to evaluate the safety and tolerability of JAB-21822 monotherapy and combination therapy in adult participants with advanced solid tumors harboring KRAS G12C mutation.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and tolerability of JAB-21822 monotherapy to determine the MTD and PR2D during Dose Escalation phase; then to evaluate preliminary antitumor activity when JAB-21822 administered alone and combination with cetuximab during Dose Expansion phase in adult participants with advanced solid tumors harboring KRAS G12C mutation.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be able to provide an archived tumor sample
* Histologically or cytologically confirmed solid tumors with KRAS G12C mutation
* Must have received at least 1 prior standard therapy
* Must have at least 1 measurable lesion per RECIST v1.1
* Must have adequate organ function
* Must be able to swallow and retain orally administered medication

Exclusion Criteria:

* Has brain or spinal metastases, except if treated and no evidence of radiographic progression or hemorrhage for at least 28 days
* Active infection requiring systemic treatment within 7 days
* Active HBV or HCV
* Any severe and/or uncontrolled medical conditions
* LVEF ≤50% assessed by ECHO or QTcF
* QT interval >470 msec
* Experiencing unresolved CTCAE 5.0 Grade >1 toxicities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
Dose Escalation phase: Number of participants with dose limiting toxicities (DLTs) | At the end of Cycle 1 (each cycle is 21 days)
Dose Escalation and Dose Expansion phase: Number of participants with adverse events | Up to 4 years
  Patients will be assessed for incidence and severity of adverse events (AEs) according to NCI-CTCAE criteria
Dose Expansion phase: Overall response rate (ORR) | Up to 4 years - from baseline to RECIST confirmed Progressive Disease
  ORR is defined as the percentage of participants with complete response (CR) or partial response (PR) per RECIST v 1.1
Dose Expansion phase: Duration of response ( DOR ) | Up to 4 years
  DOR is defined as the time from the participant's initial objective response (CR or PR) to disease progression per CTCAE v1.1 or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Dose Escalation and Dose Expansion phase: Peak Plasma Concentration (Cmax) | Up to 4 years
  Cmax of JAB-21822 alone or JAB-21822 plus cetuximabn will be measured by using plasma PK samples
Dose Escalation and Dose Expansion phase: Area under the plasma concentration versus time curve (AUC) | Up to 4 years
  AUC of JAB-21822 alone or JAB-21822 plus cetuximab will be measured by using plasma PK samples
Dose Escalation phase: Overall response rate (ORR) | Up to 4 years - from baseline to RECIST confirmed Progressive Disease
  The percentage of participants with complete response (CR) or partial response (PR) on RECIST v 1.1.
Dose Escalation phase: Duration of response ( DOR ) | Up to 4 years
  DOR is defined as the time from the participant's initial objective response (CR or PR) to disease progression per CTCAE v1.1 or death due to any cause, whichever occurs first.
Dose Escalation and Dose Expansion phase: Disease Control Rate ( DCR ) | Up to 4 years
  DCR is defined as percentage of participants with complete response (CR), partial response (PR), or stable disease(SD) per CTCAE v1.1
Dose Escalation and Dose Expansion phase: Progression-free survival (PFS) | Up to 4 years
  PFS is defined as the interval of time between the date of first treatment to the earliest date of disease progression per CTCAE v1.1 or death which occurs first

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Mayo Clinc, Phoenix, Arizona
  - Mayo Clinc, Scottsdale, Arizona
  - Mayo Clinc, Jacksonville, Florida
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Li J, Deng T, Gu Y, Calles Blanco A, Li Z, Bai C, Wu L, Huang J, Li X, Yao Y, Song Z, Li Y, Liu L, Xing L, Wu W, Martinez-Perez J, Hubert A, Zugazagoitia J, Zhang J, Wang Y, Zhao Y, Wen G, Xia G, Zhong D, Chen X, Jiang K, Wang-Gillam A, Ding Y, Liu S, Rao Z, Liu X, Shen L. Efficacy and safety of glecirasib in solid tumors with KRAS G12C mutation: A pooled analysis of two phase I/II trials. Cancer Commun (Lond). 2025 Nov;45(11):1500-1512. doi: 10.1002/cac2.70056. Epub 2025 Oct 2. PMID 41037823